CLINICAL TRIAL: NCT06522035
Title: Evaluation of Allocetra by Intra-articular Injection for the Treatment of Psoriatic Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENX-CL-06-001
Record Dates: First submitted 2024-07-07; First posted 2024-07-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 (Experimental): Stage 1 will include patients who have been treated with standard PsA therapies, and are insufficiently responsive to treatment in one or more involved joints.
  Interventions: Drug: Allocetra
- Stage 2 (Experimental): Stage 2 will include patients with oligoarticular PsA (1-4 joints involved), who have received at least one injection of corticosteroids to the target joint with insufficient response.
  Interventions: Drug: Allocetra

INTERVENTIONS:
Drug: Allocetra — Intra-articular injecton of Allocetra into the target joint.

SUMMARY:
This is an open label study to evaluate the safety and initial efficacy of intra-articular administration of Allocetra in patients with Psoriatic Arthritis (PsA).

DETAILED DESCRIPTION:
Psoriatic Arthritis (PsA) is a prevalent chronic inflammatory disease that mainly affects the synovial joints, and leads to inflammatory arthritis, in addition to skin manifestations. If left untreated, inflammatory arthritis leads to joint damage and deformities.

Allocetra is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

As macrophages play a crucial role in the initiation of PsA immunopathogenesis, they are considered an emerging target for PsA treatment.

This study will assess the safety of Allocetra injection to the joint (knee, elbow or ankle) in patients with PsA, and evaluate the preliminary responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PsA.
2. Stage 1 patients:

   At least one joint resistant to standard PsA treatments and on a stable dose of approved PsA treatment for at least 3 months prior to treatment.
3. Stage 2 patients:

   At least one symptomatic joint following attempt of intra-articular injection of corticosteroids, with insufficient response.
4. Acceptable blood tests- Complete Blood Count (CBC), electrolytes, adequate renal function, adequate liver function.

Exclusion Criteria:

1. Prior intra-articular injection to the target joint of steroids, hyaluronate or other drugs within 3 months prior to treatment.
2. Any significant injury to the target joint within the 6 months prior to treatment, or any surgery to the target joint within the 12 months prior to treatment.
3. Findings of acute fractures, severe loss of bone density, chondrocalcinosis and/or severe bone or joint deformity in the target joint.
4. Evidence of active local infection in the target joint.
5. Concomitant rheumatic, inflammatory or autoimmune disease other than PsA.
6. Other limb pain of unknown etiology.
7. Any evidence of clinically significant active infection.
8. Major medical condition as detailed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 12 months
  Number and severity of AEs, SAEs and injection reactions following treatment

SECONDARY OUTCOMES:
Patient reported pain Numeric Rating Scale (NRS) in the target joint. | 3 months, 6 months and 12 months.
  Evaluation of change from baseline in patient reported pain Numeric Rating Scale (NRS) in the target joint.

OTHER OUTCOMES:
Exploratory outcome- assessment of change from baseline in Psoriasis Area and Severity Index (PASI). | 12 months
Exploratory outcome- assessment of change from baseline in Disease Activity in Psoriatic Arthritis (DAPSA) score. | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center - Ichilov, Tel Aviv